CLINICAL TRIAL: NCT05787860
Title: Characterizing the Molecular Cutaneous Phenotype of Seborrheic Dermatitis and Treatment Response to Ruxolitinib 1.5% Cream
Brief Title: Ruxolitinib in Seborrheic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Principal Investigator, Benjamin Ungar, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 22-0672
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Seborrheic Dermatitis
MeSH Terms: conditions — Dermatitis, Seborrheic | interventions — ruxolitinib

STUDY DESIGN:
Intervention Model Description: Open-Label Trial
Masking Description: Open-Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ruxolitinib Cream (Active Comparator): Participants will receive topical ruxolitinib 1.5% cream
  Interventions: Drug: Ruxolitinib 1.5% Cream
- Healthy Control Subjects (No Intervention): Age- and gender-matched healthy control subjects

INTERVENTIONS:
Drug: Ruxolitinib 1.5% Cream — topical ruxolitinib 1.5% cream twice daily for 4 weeks
  Arms: Ruxolitinib Cream

SUMMARY:
This study is an open-label prospective interventional trial that will assess the efficacy of ruxolitinib in the treatment of seborrheic dermatitis. It will also attempt to characterize the molecular immune profiles of patients with SD at week 0 and week 4, with comparison to baseline profiles in healthy control subjects.

DETAILED DESCRIPTION:
The study will include 25 adult patients with moderate-to-severe-SD as well as 20 age- and gender-matched healthy control subjects for comparison. The SD patients will have baseline clinical score of at least 6 using the SD Severity Score in Appendix 1, or an Investigator Global Assessment (IGA) score of at least 3. Enrolled SD subjects will apply topical ruxolitinib 1.5% cream twice daily for 4 weeks. They will return for visits at weeks 2, 4, and 6 following study treatment initiation for repeat clinical assessments, medication reviews, tape-strip, blood and urine sample collections, and monitoring for adverse events.

ELIGIBILITY:
Inclusion Criteria For SD Subjects:

* Male or female subjects ≥ 18 years of age at the time of signing the informed consent document.
* Subject is able to understand and voluntarily sign an informed consent document prior to participation in any study assessments or procedures.
* Subject is able to adhere to the study visit schedule and other protocol requirements.
* Baseline SD score of IGA ≥ 3 with facial involvement
* Subject agrees to discontinue all treatments for SD from screening through study completion aside from the study drug
* Subject has failed an adequate course of treatment with at least one available therapy (topical antifungals or low-potency topical corticosteroids)
* Subject is judged to be in otherwise good overall health as judged by the investigator, based on medical history, physical examination, and laboratory testing. (NOTE: The definition of good health means a subject does not have uncontrolled significant co-morbid conditions).
* Females of childbearing potential (FCBP) must have a negative pregnancy test at Screening and Baseline. While on the study drug and for at least 90 days after the last application of the study drug, male and female participants must be willing to take appropriate contraceptive measures to avoid pregnancy or fathering a child. FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options described below:

  * Option 1: Any one of the following highly effective contraceptive methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy, OR:
  * Option 2: Male or female condom (latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]); PLUS one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.

The female subject's chosen form of contraception must be effective by the time the female subject is enrolled into the study.

Inclusion Criteria For Control Subjects:

* Male or female subjects ≥ 18 years of age at the time of signing the informed consent document.
* Subject is able to understand and voluntarily sign an informed consent document prior to participation in any study assessments or procedures.
* Subject does not currently have and does not have a history of SD.
* Female of childbearing potential (FCBP) must have a negative pregnancy test at Screening and Baseline

Exclusion Criteria For SD Subjects:

The presence of any of the following will exclude a subject from enrollment:

* SD clinical severity of IGA <3 and SD Severity Score <6.
* Subjects with other skin diseases that would interfere with the study assessment in the opinion of the investigator.
* Active bacterial, fungal, or viral skin infection within 2 weeks from study initiation.
* Subject has clinically significant (as determined by the investigator) renal, hepatic, hematologic, intestinal, endocrine, pulmonary, cardiovascular, neurological, psychiatric, immunologic, or other major uncontrolled diseases (e.g., malignancy, TB, HIV, HBV, HCV, thromboembolic events) that will affect the health of the subject during the study, or interfere with the interpretation of study results.
* Subject has previously received treatment with oral or topical JAK inhibitors
* Current other topical treatments (e.g., topical corticosteroids, topical calcineurin inhibitors) within 1 week of baseline
* Use of systemic immunosuppressive medications, including, but not limited to, cyclosporine, systemic or intralesional corticosteroids, mycophenolate mofetil, azathioprine, methotrexate, tacrolimus within 4 weeks of study initiation
* Concurrent use of strong CYP3A4 inhibitors within 7 days or 5 half-lives (whichever is longer). A list of CYP3A4 inhibiting medications can be found in Appendix 3.
* History of adverse systemic or allergic reactions to any component of the study drug.
* Current participation in any other study with an investigational medication
* Subject who is pregnant or breast feeding

Exclusion Criteria For Control Subjects:

* Active bacterial, fungal, or viral skin infection within 2 weeks from Screening/Baseline visit.
* Subject has uncontrolled clinically significant (as determined by the investigator) renal, hepatic, hematologic, intestinal, endocrine, pulmonary, cardiovascular, neurological, psychiatric, immunologic, or other disease.
* Subject has previously received treatment with oral or topical JAK inhibitors
* Current other topical treatments (e.g., topical corticosteroids, topical calcineurin inhibitors) within 1 week of baseline
* Use of systemic immunosuppressive medications, including, but not limited to, cyclosporine, systemic or intralesional corticosteroids, mycophenolate mofetil, azathioprine, methotrexate, tacrolimus within 4 weeks of study initiation
* Current participation in any other study with an investigational medication
* Subject who is pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Ungar, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Results will be provided as aggregated data.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ruxolitinib Cream | Healthy Control Subjects
Started | 25 | 20
Completed | 25 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ruxolitinib Cream | Healthy Control Subjects | Total
Number analyzed (Participants) | 25 | 20 | 45
Age, Continuous [Mean (Full Range); unit: years] | 46 [23 to 72] | 42 [21 to 71] | 45 [21 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 17 | 10 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 9 | 20
  Not Hispanic or Latino | 14 | 11 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 3 | 12
  White | 14 | 15 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Investigator Global Assessment of 0 or 1 at Week 4
Description: Number of Participants with Investigator Global Assessment of 0 or 1 at Week 4
  IGA Scale from 0-4
  Clear 0 No signs of SD
  Almost Clear 1 Just perceptible erythema and just perceptible scaling
  Mild 2 Mild erythema and mild scaling
  Moderate 3 Moderate erythema and moderate scaling
  Severe 4 Severe erythema and severe scaling
Time Frame: At end of Treatment, Week 4
Population: Data collected only for participants with SD
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib Cream | Healthy Control Subjects
Number analyzed (Participants) | 25 | 0
Participants | 20 |

2. Secondary Outcome: Change in Investigator Global Assessment From Baseline to Week 4
Description: IGA Scale from 0-4
  Clear 0 No signs of SD
  Almost Clear 1 Just perceptible erythema and just perceptible scaling
  Mild 2 Mild erythema and mild scaling
  Moderate 3 Moderate erythema and moderate scaling
  Severe 4 Severe erythema and severe scaling
Time Frame: Baseline and Week 4
Population: Data collected only for participants with SD
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ruxolitinib Cream | Healthy Control Subjects
Number analyzed (Participants) | 25 | 0
score on a scale | -2.16 (0.69) |

3. Secondary Outcome: Mean Change in Seborrheic Dermatitis Severity Score
Description: Mean Change in seborrheic dermatitis severity score from baseline and week 4, baseline a d week 6 and week 4 and week 6
  SD Severity Score (the sum of the three clinical features for a total score ranging from 0-12), where higher scores indicate more severe outcomes.
  Scale 0-4 Erythema 0-4 Pruritus 0-4 (0 = absence, 1 = mild, 2 = moderate, 3 = significant, 4 = severe)
Time Frame: Baseline, Week 4, Week 6
Population: Data collected only for participants with SD
Measure: Mean (Standard Deviation); unit: mean change in score on a scale
Arm/Group | Ruxolitinib Cream | Healthy Control Subjects
Number analyzed (Participants) | 25 | 0
mean change in score on a scale
  baseline and week 4 | -6 (1.61) |
  baseline and week 6 | -2.8 (2.96) |
  week 4 and week 6 | 3.2 (2.52) |

4. Secondary Outcome: Mean Change in Seborrheic Dermatitis Severity Score for Scale
Description: Mean Change in seborrheic dermatitis severity score for Scale from baseline and week 4, baseline and week 6, week 4 and week 6
  Scale 0-4, where higher scores indicate more severe outcomes.
  (0 = absence, 1 = mild, 2 = moderate, 3 = significant, 4 = severe)
Time Frame: Baseline, Week 4, and Week 6
Population: Data collected only for participants with SD
Measure: Mean (Standard Deviation); unit: mean change in score on a scale
Arm/Group | Ruxolitinib Cream | Healthy Control Subjects
Number analyzed (Participants) | 25 | 0
mean change in score on a scale
  baseline and week 4 | -1.56 (0.87) |
  baseline and week 6 | -0.56 (1.29) |
  week 4 and week 6 | 3.2 (2.52) |

5. Secondary Outcome: Change in Seborrheic Dermatitis Severity Score for Erythema
Description: Change in seborrheic dermatitis severity score for Erythema from baseline and week 4, baseline and week 6, week 4 and week 6
  Erythema 0-4, where higher scores indicate more severe outcomes.
  (0 = absence, 1 = mild, 2 = moderate, 3 = significant, 4 = severe)
Time Frame: Baseline, Week 4, and Week 6
Population: Data collected only for participants with SD
Measure: Mean (Standard Deviation); unit: mean change in score on a scale
Arm/Group | Ruxolitinib Cream | Healthy Control Subjects
Number analyzed (Participants) | 25 | 0
mean change in score on a scale
  baseline and week 4 | -2 (0.76) |
  baseline and week 6 | -1.04 (1.06) |
  week 4 and week 6 | 0.96 (0.98) |

6. Secondary Outcome: Change in Seborrheic Dermatitis Severity Score for Pruritus
Description: Change in seborrheic dermatitis severity score for Pruritus from baseline and week 4, baseline and week 6, week 4 and week 6
  Pruritus 0-4, where higher scores indicate more severe outcomes.
  (0 = absence, 1 = mild, 2 = moderate, 3 = significant, 4 = severe)
Time Frame: Baseline Week 4, and Week 6
Population: Data collected only for participants with SD
Measure: Mean (Standard Deviation); unit: mean change in score on a scale
Arm/Group | Ruxolitinib Cream | Healthy Control Subjects
Number analyzed (Participants) | 25 | 0
mean change in score on a scale
  baseline and week 4 | -2.44 (0.71) |
  baseline and week 6 | -1.2 (1.12) |
  week 4 and week 6 | 1.24 (0.97) |

7. Secondary Outcome: Frequency of Adverse Events
Time Frame: 6 weeks
Measure: Number; unit: events
Arm/Group | Ruxolitinib Cream | Healthy Control Subjects
Number analyzed (Participants) | 25 | 20
events | 0 | 0

8. Secondary Outcome: Duration of Adverse Events
Time Frame: 6 weeks
Population: As there were no adverse events, duration could not be calculated.
Arm/Group | Ruxolitinib Cream | Healthy Control Subjects
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Severity of Adverse Events
Description: Severity will be measured as a category (mild, moderate, or severe).
Time Frame: 6 weeks
Population: As there were no adverse events, severity of adverse events could not be calculated.
Arm/Group | Ruxolitinib Cream | Healthy Control Subjects
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Ruxolitinib Cream | Healthy Control Subjects
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/20
Other Adverse Events (participants affected / at risk) | 0/25 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-02): https://cdn.clinicaltrials.gov/large-docs/60/NCT05787860/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-28): https://cdn.clinicaltrials.gov/large-docs/60/NCT05787860/ICF_001.pdf